CLINICAL TRIAL: NCT00773305
Title: Chart Review of the Efficacy of Prostate Seed Implantation for Local Control of Early Stage Prostate Cancer
Brief Title: Efficacy of Prostate Seed Implantation for Local Control of Early Stage Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Summa Health System (Other)
Responsible Party: Principal Investigator, William Demas, Study Principal Investigator, Summa Health System
Other Study IDs: Prostate Seed Implantation
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2012-12-28 (Estimated); Status verified 2012-12

CONDITIONS: Prostate Cancer
Keywords: seed implantation
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary goal of this project is to evaluate the efficacy of prostate seed implantation for the treatment of early stage prostate cancer for patients treated at Summa Health System/Akron City Hospital and Salem Community Hospital.

DETAILED DESCRIPTION:
Charts of early stage prostate cancer patients receiving prostate seed implants with or without external beam radiotherapy and/or hormonal therapy will be reviewed and abstracted. The abstracted data will include pathology reports including Gleason score and T stage, PSA, treatment assignment and dosimetry parameters including dose and percent compliant with established criteria based on guidelines established by the American Brachytherapy Society.

A database will be developed for capture of the abstracted data. Outcomes will be determined based on PSA levels at 2 and 5 years after prostate seed implantation. The role of hormonal therapy with prostate seed implantation and outcomes will be evaluated. The outcomes will be compared to national statistics.

ELIGIBILITY:
Inclusion Criteria:

* Prostate seed implantation for the treatment of early stage prostate cancer

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prostate seed implantation for the treatment of early stage prostate cancer
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2008-10; Primary Completion 2010-11 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy of prostate brachytherapy for local control of early stage prostate cancer at Summa Health System | Pre-op through 4 follow-up visits
  A retrospective chart review of PSA values on 85 patients from 2001-2008 with prostate cancer stage T1c-T2a NX MO, who were treated with permanent prostate brachytherapy using conventional transrectal ultrasound guided placement of Iodine-125 seeds delivering 145 Gy or 110 Gy, depending on whether mono or combination therapy with external beam radiotherapy (EBRT) was used. Those who had EBRT received 45 Gy prior to seed implants. Some patients also received hormonal therapy.

CONTACTS AND LOCATIONS:
Overall Officials: William Demas, MD, Principal Investigator — Summa Health System